CLINICAL TRIAL: NCT03228576
Title: Observationnal Multicenter Study on a Prospective Cohort of Kidney Transplanted Patients Receiving a Year After Transplant an Extended Releasing Tacrolimus-Everolimus Association
Brief Title: Prospective Cohort of Kidney Transplanted Patients Receiving an Extended Releasing Tacrolimus-Everolimus Association
Status: Terminated | Type: Observational
Why Stopped: No recruitment
Sponsor: Poitiers University Hospital (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: TREVISE
Record Dates: First submitted 2017-06-23; First posted 2017-07-25 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Kidney Transplant; Immunosuppression
Keywords: Tacrolimus; Envarsus; Everolimus; kidney; Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TREVISE
  Interventions: Combination Product: Extended release Tacrolimus-Everolimus association

INTERVENTIONS:
Combination Product: Extended release Tacrolimus-Everolimus association — Envarsus® will be used as Tacrolimus Certican® will be used as Everolimus

SUMMARY:
The tacrolimus-Everolimus association is used as an immunospressive treatment after a kidney transplant. It combined immunosupressive properties of both products and reduce the nephrotoxicity of tacrolimus by lowering the dosage.

The commercialisation of a new extended release Tacrolimus pharmaceutical form and the lack of information justify a modality of use and tolerence evaluation of this new association, commonly used.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients informed and giving his agreement to the use of every collected data
* Patients with kidney transplantation for at least one year and being treated with the immunosppressive assiociation of Tacrolimus (Prograf ®)-Everolimus
* Patients whose investigators decides to switch from Prograf ® to an Envarsus ®-Everolimus association

Exclusion Criteria:

* Other transplantation
* Drug or alcohol abuse
* Patients unable to understand the purpose or modalities of this study, unable to give his agreement or unable to stick to the protocol
* Patients on an interventionnal protocol when included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old with kidney transplantation for at least one year.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Tolerance of the Certican®-Envarsus® association | During 1 year, between each visit (J0, M3, M6, M9, M12)
  Assess clinical and biological tolerance of the Certican®-Envarsus® association on kidney transplanted patient, one year after transplant : study of adverse events with biological results (biochimy, hematology).
  Study of incidence of Treatment-Emergent Adverse Events.

SECONDARY OUTCOMES:
Patients description | 1 year
  Describe the profil of included patients
clinical evolution | 1 year
  Describe the patients clinical evolution after a one year follow up : adverse events, renal function (creatinine)...
Treatment | 1 year
  Describe treatments and switch modalities : tolerability with adverse events, conversion value between Prograf® and Envarsus®
Renal function | 1 year
  Describe the evolution of renal function during follow up : creatinine value during the study
Graft Rejections and survival rates | 1 year
  Assess acute graft rejections (confirmed by a biopsy with the Banff classification and creatinine value) and transplants survival rates a year after the switch : all renal biopsies will be reported, with the reason for the biopsy.
Medication compliance | 1 year
  Assess medication compliance during the switch and by the end of the study, to evaluated by doctor by asking the patient and with pharmacological concentrations (used in nephrology)

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Amiens University Hospital, Amiens
  - Angers University Hospital, Angers
  - Caen University Hospital, Caen
  - Clermont Ferrand University Hospital, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Rennes University Hospital, Rennes
  - Rouen University Hospital, Rouen
  - Strasbourg University Hospital, Strasbourg
  - Tours University Hospital, Tours